CLINICAL TRIAL: NCT00275613
Title: Pilot Study of Rituximab for Membranoproliferative Glomerulonephritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John Dillon, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 976-05
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Glomerulonephritis, Membranoproliferative
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab, IV infusion (Experimental): The Rituximab dose is 1000 mg (1 gm) given as an IV infusion every two weeks for 2 doses (days 1 and 15)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — The Rituximab dose is 1000 mg (1 gm) given as an IV infusion every two weeks for 2 doses (days 1 and 15)
  Other Names: Rituxan

SUMMARY:
Membranoproliferative glomerulonephritis (MPGN) is a relatively-rare, immune-mediated kidney disease. All current therapies are inadequate and MPGN frequently leads to kidney failure. This study is a 10 patient trial of the monoclonal antibody rituximab for adult patients with MPGN. Study patients will receive 2 doses of rituximab intravenously on days 1 and 15 and will then be followed for 1 year.

DETAILED DESCRIPTION:
Membranoproliferative glomerulonephritis (MPGN) is a relatively-rare, immune-mediated glomerular disease. There is no accepted therapy and all current therapies are inadequate. Current therapeutic options include immunosuppression with corticosteroids alone or in combination with alkylating agents, antiplatelet therapy with aspirin and/or dipyridamole and/or warfarin, and angiotensin converting enzyme inhibitors and/or angiotensin receptor blockers. As with other glomerular diseases the amount of protein in the urine correlates well with the long-term prognosis. Thus, this parameter has been used in previous studies, and will be used in this study, as the primary indicator of therapeutic efficacy. We propose a pilot study to test the hypothesis that selective B lymphocyte depletion will result in disappearance of pathogenic antibodies and induce remission of proteinuria in patients with idiopathic membranoproliferative glomerulonephritis. Our population will be 10 adults with MPGN involving either the native kidneys or a renal transplant. We will enroll patients with a glomerular filtration rate (GFR) greater than or equal to 25 ml/min, as estimated by creatinine clearance, and with a 24 hour urinary ratio of protein to creatinine greater than or equal to 1, while receiving an angiotensin converting enzyme inhibitor (ACEI) or angiotensin II receptor blocker (ARB). Patients will receive Rituximab 1g on Day 1 and 15. Patients will be followed for 1 year following completion of treatment. The primary outcome will be the change in urinary protein excretion at 6 months. Secondary outcomes will include changes in the GFR, changes in urinary protein excretion at 3, 9, and 12 months, the rate of change in urinary protein excretion, serum albumin concentration, serum cholesterol, the number of complete and partial remissions, time to remission, and the number of relapses.

ELIGIBILITY:
Inclusion Criteria:

* MPGN either native/renal transplant kidneys with biopsy last 3 years
* Age > 18 years
* Urinary protein to creatinine ratio > 1.0 in a 24-hour urine collection, despite ACE inhibitor/ARB treatment
* Patients need to be treated with an ACEI and/or ARB, for at least 3 months prior to enrollment with the systolic blood pressure < 140 mm Hg for at least 75% of readings. Goal systolic blood pressure will be < 130 mm Hg.)
* Women must be post-menopausal, surgically sterile or practicing a medically approved method of contraception
* Patients intolerant of ACE inhibitors/ARBs may enter the study without being treated with these agents
* Able/willing to give written informed consent/comply with the requirements of study protocol
* Estimated GFR ≥ 25 ml/min per 1.73m^2 in the presence of ACE inhibitor/ARB therapy. The GFR will be estimated using the 4 variable Modification of Diet in Renal Disease (MDRD) equation/National Kidney Foundation - Chronic Kidney Disease (NKF-CKD) guidelines
* Adequate liver function, indicated by bilirubin, aspartate aminotransferase (AST), and alkaline phosphatase levels not more than 2.5 times the upper normal limit
* Negative serum pregnancy test (for women of child bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment

Exclusion Criteria:

* Age <18 years.
* Estimated GFR < 25 ml/min per 1.73 m^2
* Concurrent use of immunosuppressive therapy with the exceptions of prednisone 10 mg/day or less or an equivalent amount of another glucocorticoid or, among transplant patients, stable or decreasing transplant immunosuppression. Patient must be off immunosuppressive medications for > 3 months prior to enrollment into the study
* Medical conditions causing MPGN (e.g. HIV, hepatitis B, hepatitis C, systemic lupus erythematosus, monoclonal gammopathies). Patients with idiopathic cryoglobulinemia will not be excluded
* Presence or suspicion of active infection
* Type 1 or type 2 diabetes mellitus
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous Treatment with Rituximab (MabThera®/Rituxan®) or another B-cell depleting antibody
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Human immunodeficiency virus (HIV)
* Hepatitis B or C
* History of recurrent significant or recurrent bacterial infections
* Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Ongoing use of high dose steroids(> 10 mg/day)or unstable steroid dose past 4 weeks
* Lack of peripheral venous access
* Drug,alcohol or chemical abuse within 6 months prior to screening
* Pregnancy(negative serum pregnancy test performed all women of childbearing potential within 7 days of treatment)
* Lactation
* Concomitant malignancies/previous malignancies within last 5 years, with the exception of adequately treated basal/squamous cell carcinoma of skin or carcinoma of cervix
* Major psychiatric disorder
* Significant cardiac or pulmonary disease
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory suspicion of a disease/condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Inability to comply with study and follow-up procedures

Laboratory Exclusion Criteria (Screening):

* Hemoglobin:< 8.5 gm/dL
* Platelets:< 100,000/mm
* Total bilirubin,AST/alkaline phosphatase > 2.5 x Upper Limit of Normal unless related to primary disease
* Positive Hepatitis B or C serology
* Positive HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Proteinuria | The primary endpoints are based on quantitative changes in urine protein measured at 6 months. Additional evaluations of urine protein will be done at 3, 9, and 12 months.
  1. Complete remission (CR) UP ≤ 0.3 g, without doubling of serum creatinine
  2. Partial remission (PR) Reduction in UP of > 50% plus final UP ≤ 3.5 g but >0.3 g, without doubling of serum creatinine
  3. Limited response (LR) Reduction in UP of > 50% with final UP > 3.5 g, without doubling of serum creatinine
  4. Non-response (NR) Reduction in UP of < 50%. (includes progression of UP), without doubling of serum creatinine
  5. Progression Proteinuria increases by > 50% or serum creatinine doubles
  6. Relapse New development of nephrotic range proteinuria, i.e. > 3.5 g/day

SECONDARY OUTCOMES:
Serum albumin | 3, 6, 9 and 12 months
  Change in serum albumin concentration
Serum cholesterol | 6 and 9 month timepoints
  Change in serum cholesterol levels

CONTACTS AND LOCATIONS:
Overall Officials: John J. Dillon, M.D., M.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States